CLINICAL TRIAL: NCT05777720
Title: A Cluster-randomized Controlled Trial of Air Filtration and Ventilation Improvements to Reduce SARS CoV 2 Transmission Among Household Contacts
Brief Title: Cluster-Randomized Trial of Air Filtration and Ventilation to Reduce Covid19 Spread in Homes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Abraar Karan, Post-Doctoral Fellow, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 55479; 5T32AI052073-17 (NIH)
Record Dates: First submitted 2023-03-18; First posted 2023-03-21 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Covid19
Keywords: ventilation; air filtration; Covid19; SARS CoV 2; household transmission
MeSH Terms: conditions — COVID-19; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention will be administered in this arm. Investigators will give families a CO2 monitor to measure average CO2 levels in the home. Investigators will provide a link to the basic CDC isolation guidelines which would be part of standard of care. Investigators will test family members at day 0-1 for baseline testing; and again on day 7 for assessing secondary transmission among susceptible contacts.
- Intervention (Experimental): Families are provided with one filtration fan unit per room in their home (and one for the index case; if the family lives in a studio, they would receive 2 units). Investigators will advise families on ventilation improvements in their home. Investigators will provide an instructional pamphlet that describes how the fans work and the importance of ventilation. Investigators will follow-up on day 3-4 to check in and run through a checklist to ensure the fans are working and ventilation improvements are being attempted. Investigators will give families a CO2 monitor to measure average CO2 levels in the home. Investigators will test family members at day 0-1 for baseline testing; and again on day 7 for assessing secondary transmission among susceptible contacts.
  Interventions: Device: Filtration Fan; Behavioral: Safe-home pamphlet; Behavioral: Mid-week phone call

INTERVENTIONS:
Device: Filtration Fan — Investigators are using box fans with attached MERV16 filters, a design that has been tested and published in the scientific literature.
  Arms: Intervention
Behavioral: Safe-home pamphlet — The pamphlet has information on how the filtration fans work through visual images; and images of ventilation improvements in the home through opening windows.
  Arms: Intervention
Behavioral: Mid-week phone call — On day 3-4 of the study, the study coordinator assigned to the house will call and check in regarding the filtration fan usage and remind families about the importance of filtration and ventilation.
  Arms: Intervention

SUMMARY:
Investigators are evaluating whether an intervention consisting of box-fans with MERV 16 filters ("filtration fans") and recommendations for improving ventilation in the home can reduce secondary spread of Covid19 from an index case to susceptible contacts within the home.

ELIGIBILITY:
Inclusion Criteria:

* Household members live in a shared space (apartment, home) with others (as opposed to renting single rooms in a shared space, for example)
* At least 3 other people live in the household aside from index case

Exclusion Criteria:

* If index case test positive day was over 2 days prior
* If half or more household members are thought to be infected already
* If household has fewer than 3 contacts interested in participating in the study
* If fewer than 3 contacts are expected to be present in the house for a majority of the following 7 days

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Covid19 | 7th day since enrollment in the trial
  Investigators will measure the incidence of Covid19 in susceptible contacts on day 7.

SECONDARY OUTCOMES:
Incidence of new upper respiratory symptoms | 7th day since enrollment in the trial
  Investigators will measure reported new upper respiratory symptoms in susceptible contacts.
Average CO2 levels | 7 days
  Investigators will measure 7 day average CO2 levels in the home (measured in parts per million)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Maldonado, MD, Study Director — Stanford University; Abraar Karan, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - San Mateo Medical Center, San Mateo, California
  - Stanford University Medical Center, Stanford, California

IPD SHARING:
Plan to Share IPD: No